CLINICAL TRIAL: NCT00057863
Title: A Phase II Study of Oxaliplatin in Combination With Paclitaxel in Patients With Locally Recurrent or Metastatic Cervical Cancer
Brief Title: Oxaliplatin and Paclitaxel in Treating Patients With Locally Recurrent or Metastatic Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03004; NCI-2012-03004 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-5840; 0902-492 (Other: Montefiore Medical Center - Moses Campus); 5840 (Other: CTEP); N01CM62204 (NIH); P30CA013330 (NIH)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2012-12

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma; Recurrent Cervical Carcinoma; Stage IVA Cervical Cancer; Stage IVB Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Taxes; Oxaliplatin

ARMS (1):
- Treatment (paclitaxel, oxaliplatin) (Experimental): Patients receive paclitaxel IV over 3 hours and oxaliplatin IV over 2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; TAX
Drug: Oxaliplatin — Given IV

SUMMARY:
Phase II trial to study the effectiveness of combining oxaliplatin with paclitaxel in treating patients who have locally recurrent or metastatic cervical cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rates for the combination of paclitaxel and oxaliplatin in patients with metastatic or locally recurrent cervical cancer.

II. To determine the toxicities and recovery from toxicities of patients with cervical cancer receiving paclitaxel and oxaliplatin.

OUTLINE:

Patients receive paclitaxel IV over 3 hours and oxaliplatin IV over 2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed ever 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed squamous cell, adenosquamous cell or adenocarcinoma of the uterine cervix
* Lesions must be metastatic to organs or lymph nodes outside the pelvis or must be locally recurrent in the pelvis after definitive therapy (surgery or radiation therapy) with at least 50% increase in size on sequential imaging studies
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Patients may have received chemotherapy in conjunction with radiation therapy for primary, definitive therapy; patients may not have received treatment with cytotoxic agents for advanced or recurrent disease
* Patients who have had chemotherapy, radiation therapy or surgery must allow four weeks for recovery of bone marrow or recovery from surgery/radiation
* Life expectancy of greater than 2 months
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits
* The effects of oxaliplatin on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to oxaliplatin, cisplatin or carboplatin or paclitaxel or docetaxel
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because oxaliplatin is a platinating agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with oxaliplatin and paclitaxel, breastfeeding should be discontinued if the mother is treated with oxaliplatin
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with oxaliplatin or other agents administered during the study; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2003-01; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Kuo, Principal Investigator — Montefiore Medical Center - Moses Campus
Locations (1):
- Montefiore Medical Center - Moses Campus, The Bronx, New York, United States

REFERENCES:
- [Derived] Kuo DY, Blank SV, Christos PJ, Kim M, Caputo TA, Pothuri B, Hershman D, Goldman N, Ivy PS, Runowicz CD, Muggia F, Goldberg GL, Einstein MH. Paclitaxel plus oxaliplatin for recurrent or metastatic cervical cancer: a New York Cancer Consortium Study. Gynecol Oncol. 2010 Mar;116(3):442-6. doi: 10.1016/j.ygyno.2009.10.082. Epub 2009 Nov 20. PMID 19931137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 35 patients were enrolled in the study from April 2003 until August 2008.
Period: Overall Study
Arm/Group | Treatment (Paclitaxel, Oxaliplatin)
Started | 35
Completed | 32
Not Completed | 3
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Paclitaxel, Oxaliplatin)
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 56 [27 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 12
  Hispanic | 9
  Black | 8
  Asian | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response Rate (CR+PR)
Description: 95% confidence interval will be estimated via binomial proportions.
Time Frame: Up to 7 years
Measure: Number; unit: participants
Arm/Group | Treatment (Paclitaxel, Oxaliplatin)
Number analyzed (Participants) | 32
participants
  Complete Response | 2
  Partial Respone | 5
  Stable disease | 8

2. Secondary Outcome: Progression-free Survival
Description: Assessed by Kaplan-Meier survival analysis and 95% confidence intervals will be calculated using Greenwood's formulae.
Time Frame: From first treatment day until objective or symptomatic progression or death, assessed up to 7 years
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | Treatment (Paclitaxel, Oxaliplatin)
Number analyzed (Participants) | 32
weeks | 21 [14.7 to 27.2]

3. Secondary Outcome: Overall Survival
Description: Assessed by Kaplan-Meier survival analysis and 95% confidence intervals will be calculated using Greenwood's formulae.
Time Frame: From first treatment day until death, assessed up to 7 years
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | Treatment (Paclitaxel, Oxaliplatin)
Number analyzed (Participants) | 32
weeks | 52 [39.4 to 64.8]

4. Secondary Outcome: Toxicities, Assessed and Graded According to CTCAE Version 3.0
Description: Exact 95% confidence intervals will be calculated. The 95% confidence interval was not calculated for the toxicities
Time Frame: Up to 7 years
Population: There were 135 cycles administered.
Measure: Number; unit: percentage of grade 3/4
Arm/Group | Treatment (Paclitaxel, Oxaliplatin)
Number analyzed (Participants) | 32
percentage of grade 3/4
  grade 3/4 hematologic toxicities | 20.1
  grade 3/4 non-hematologic toxicities | 34.1

ADVERSE EVENTS:
Arm/Group | Treatment (Paclitaxel, Oxaliplatin)
Serious Adverse Events (participants affected / at risk) | 32/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Paclitaxel, Oxaliplatin) (N=32)
Neutropenia (Blood and lymphatic system disorders) | 8 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 12 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Thrombosis (Vascular disorders) | 2 (2)
Coagulopathy (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Severe vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Bowel perforation fistula (Gastrointestinal disorders) | 3 (3)
Neuropathy (Nervous system disorders) | 5 (5)
Pain (General disorders) | 8 (8)
Weakness (General disorders) | 5 (5)
Electrolytes imbalance (Metabolism and nutrition disorders) | 14 (14)
Dehydration (Gastrointestinal disorders) | 1 (1)
Hypersensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Psychological (Psychiatric disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Death NOS (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Paclitaxel, Oxaliplatin) (N=32)
Fatigue (General disorders) | 9 (9)
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8)
Pain: back (Musculoskeletal and connective tissue disorders) | 2 (2)
Edema:limb (General disorders) | 3 (3)
Leukocytes (Investigations) | 5 (5)
Pain: Bone (Musculoskeletal and connective tissue disorders) | 2 (2)
Fever (General disorders) | 3 (3)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 2 (2)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2)
Pain: Abdomen (Gastrointestinal disorders) | 2 (2)
Pain: Joint (Musculoskeletal and connective tissue disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Ataxia (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less